CLINICAL TRIAL: NCT00105716
Title: Study to Lower Veterans Blood Pressure: Patient/Physician Intervention
Brief Title: Study to Lower Veterans BP: Patient/Physician Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IIR 20-034
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-04

CONDITIONS: Hypertension
Keywords: hypertension; adherence; cardiovascular diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telephone behavioral education; Behavioral: Computer behavioral education

INTERVENTIONS:
Behavioral: Telephone behavioral education
Behavioral: Computer behavioral education

SUMMARY:
This four and a half year trial is evaluating both a patient and a provider intervention in a primary care setting among diagnosed hypertensive veterans. The two primary hypotheses are: 1) the proportion of veterans with BP control who receive either the provider-directed decision support or the patient health education and behavioral intervention will be increased by 10% as compared to usual care; and 2) the proportion of veterans with BP control who receive both the provider-directed decision support and the patient health education and behavioral intervention will be increased by 25% as compared to usual care.

DETAILED DESCRIPTION:
Background:

There are 65 million Americans and over 8.5 million veterans who have been diagnosed with hypertension, yet only 31% have their blood pressure (BP) under effective control. Uncontrolled hypertension greatly increases the risk of stroke, CAD, renal failure, CHF, and mortality.

Objectives:

This four year study evaluated simultaneously both a patient and a provider intervention in a primary care setting among diagnosed hypertensive veterans. The two primary hypotheses were: 1) the proportion of veterans with BP control who receive either the provider-directed decision support or the patient behavioral/education intervention will be increased by 10% as compared to usual care; and 2) the proportion of veterans with BP control who receive both the provider-directed decision support and the patient health education and behavioral intervention will be increased by 25% as compared to usual care.

Methods:

This was a randomized controlled trial with a split-plot design. Thirty primary care providers in the Durham VAMC Primary Care Clinic were randomly assigned to receive either the provider intervention or basic patient information; 588 of their hypertensive patients were randomized to the patient intervention or usual care. The provider intervention (ATHENA study (IIR 99-275) included an electronically generated hypertension decision support system (DSS) delivered to the provider at each hypertensive patient's visit. The provider intervention was designed to improve guideline concordant therapy. The patient intervention was a tailored behavioral/education intervention administered at periodic telephone contacts. The intervention included support and reminders, information on hypertension and on health behaviors. Patients received feedback about their recent BP values, continuous patient education, and were monitored and supported to enhance adherence. The control group was usual care.

Status:

Complete. Major activities completed in the past 12 months include submission of a manuscript describing the study, the interventions, and baseline and follow-up analyses. Secondary analyses are being completed which will be included in additional manuscripts.

ELIGIBILITY:
Inclusion Criteria:

1. >1 ICD9 Diagnosis 401.0, 401.1, 401.9
2. Designated Primary Care Provider
3. >1 Primary Care visit between 1/01/01-12/31/01
4. Restricted to NC and VA addresses
5. >1 Medication CV100, CV150, CV200, CV490, CV701, CV702, CV704, CV800, CV805

Exclusion Criteria:

1. Dialysis patient
2. Hospitalization for stroke in prior 3 months
3. Myocardial infarction in prior 3 months
4. Coronary artery revascularization in prior 3 months
5. Metastatic cancer diagnosis in prior 3 months
6. Transplant of: kidney; liver; lung; pancreas; peripheral stem cells; bone; bone marrow; heart; intestine; stem cells; tissue V42.9; complications of transplants
7. Nursing home resident
8. Documented diagnosis of dementia
9. Difficulty hearing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2002-03; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
BP control at primary care visit; Systolic and diastolic BPs as recorded at each primary care provider visit during 24 month enrollment period.

SECONDARY OUTCOMES:
Knowledge and perceived risks associated with hypertension and ability to continue hypertension regimen will be assessed at baseline and via telephone 6 and 24 months after baseline; Medication adherence will be assessed from pharmacy records

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B. Bosworth, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Eugene Z. Oddone, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Datta SK, Oddone EZ, Olsen MK, Orr M, McCant F, Gentry P, Bosworth HB. Economic analysis of a tailored behavioral intervention to improve blood pressure control for primary care patients. Am Heart J. 2010 Aug;160(2):257-63. doi: 10.1016/j.ahj.2010.05.024. PMID 20691830
- [Result] Powers BJ, Olsen MK, Oddone EZ, Bosworth HB. The effect of a hypertension self-management intervention on diabetes and cholesterol control. Am J Med. 2009 Jul;122(7):639-46. doi: 10.1016/j.amjmed.2008.12.022. PMID 19559166
- [Result] Thorpe CT, Bryson CL, Maciejewski ML, Bosworth HB. Medication acquisition and self-reported adherence in veterans with hypertension. Med Care. 2009 Apr;47(4):474-81. doi: 10.1097/mlr.0b013e31818e7d4d. PMID 19330891
- [Result] Bosworth HB, Olsen MK, Dudley T, Orr M, Goldstein MK, Datta SK, McCant F, Gentry P, Simel DL, Oddone EZ. Patient education and provider decision support to control blood pressure in primary care: a cluster randomized trial. Am Heart J. 2009 Mar;157(3):450-6. doi: 10.1016/j.ahj.2008.11.003. Epub 2009 Jan 10. PMID 19249414
- [Result] Powers BJ, Olsen MK, Oddone EZ, Thorpe CT, Bosworth HB. Literacy and blood pressure--do healthcare systems influence this relationship? A cross-sectional study. BMC Health Serv Res. 2008 Oct 23;8:219. doi: 10.1186/1472-6963-8-219. PMID 18947408
- [Result] Olsen MK, DeLong ER, Oddone EZ, Bosworth HB. Strategies for analyzing multilevel cluster-randomized studies with binary outcomes collected at varying intervals of time. Stat Med. 2008 Dec 20;27(29):6055-71. doi: 10.1002/sim.3446. PMID 18825655
- [Result] Walsh JM, Sundaram V, McDonald K, Owens DK, Goldstein MK. Implementing effective hypertension quality improvement strategies: barriers and potential solutions. J Clin Hypertens (Greenwich). 2008 Apr;10(4):311-6. doi: 10.1111/j.1751-7176.2008.07425.x. PMID 18401229
- [Result] Cho AH, Voils CI, Yancy WS Jr, Oddone EZ, Bosworth HB. Does participatory decision making improve hypertension self-care behaviors and outcomes? J Clin Hypertens (Greenwich). 2007 May;9(5):330-6. doi: 10.1111/j.1524-6175.2007.06489.x. PMID 17485968
- [Result] Powers BJ, Oddone EZ, Grubber JM, Olsen MK, Bosworth HB. Perceived and actual stroke risk among men with hypertension. J Clin Hypertens (Greenwich). 2008 Apr;10(4):287-94. doi: 10.1111/j.1751-7176.2008.07797.x. PMID 18401226
- [Result] Lin ND, Martins SB, Chan AS, Coleman RW, Bosworth HB, Oddone EZ, Shankar RD, Musen MA, Hoffman BB, Goldstein MK. Identifying barriers to hypertension guideline adherence using clinician feedback at the point of care. AMIA Annu Symp Proc. 2006;2006:494-8. PMID 17238390
- [Result] Lowry KP, Dudley TK, Oddone EZ, Bosworth HB. Intentional and unintentional nonadherence to antihypertensive medication. Ann Pharmacother. 2005 Jul-Aug;39(7-8):1198-203. doi: 10.1345/aph.1E594. Epub 2005 Jun 14. PMID 15956238
- [Result] Bosworth HB, Olsen MK, Goldstein MK, Orr M, Dudley T, McCant F, Gentry P, Oddone EZ. The veterans' study to improve the control of hypertension (V-STITCH): design and methodology. Contemp Clin Trials. 2005 Apr;26(2):155-68. doi: 10.1016/j.cct.2004.12.006. PMID 15837438
- [Result] Bosworth HB, Oddone EZ. A model of psychosocial and cultural antecedents of blood pressure control. J Natl Med Assoc. 2002 Apr;94(4):236-48. PMID 11991336
- [Result] Chan AS, Coleman RW, Martins SB, Advani A, Musen MA, Bosworth HB, Oddone EZ, Shlipak MG, Hoffman BB, Goldstein MK. Evaluating provider adherence in a trial of a guideline-based decision support system for hypertension. Stud Health Technol Inform. 2004;107(Pt 1):125-9. PMID 15360788
- [Result] Steinman MA, Fischer MA, Shlipak MG, Bosworth HB, Oddone EZ, Hoffman BB, Goldstein MK. Clinician awareness of adherence to hypertension guidelines. Am J Med. 2004 Nov 15;117(10):747-54. doi: 10.1016/j.amjmed.2004.03.035. PMID 15541324
- [Result] Bosworth HB, Dudley T, Olsen MK, Voils CI, Powers B, Goldstein MK, Oddone EZ. Racial differences in blood pressure control: potential explanatory factors. Am J Med. 2006 Jan;119(1):70.e9-15. doi: 10.1016/j.amjmed.2005.08.019. PMID 16431192
- [Result] Hong TB, Oddone EZ, Dudley TK, Bosworth HB. Subjective and objective evaluations of health among middle-aged and older veterans with hypertension. J Aging Health. 2005 Oct;17(5):592-608. doi: 10.1177/0898264305279780. PMID 16177452
- [Result] Bosworth HB, Olsen MK, Gentry P, Orr M, Dudley T, McCant F, Oddone EZ. Nurse administered telephone intervention for blood pressure control: a patient-tailored multifactorial intervention. Patient Educ Couns. 2005 Apr;57(1):5-14. doi: 10.1016/j.pec.2004.03.011. PMID 15797147